CLINICAL TRIAL: NCT03003728
Title: 2015-10: A Phase II Pilot Study of Expanded Natural Killer Cells and Elotuzumab to Eradicate High-Risk Myeloma Post Autologous Stem Cell Transplant
Brief Title: 2015-10: Expanded Natural Killer Cells and Elotuzumab for High-Risk Myeloma Post- Autologous Stem Cell Transplant (ASCT)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawal of study support
Sponsor: University of Arkansas (Other)
Collaborators: Bristol-Myers Squibb (Industry); Altor BioScience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205009
Record Dates: First submitted 2016-12-21; First posted 2016-12-28 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; Melphalan; Cell Count; ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Treatment (Experimental): Elotuzumab 10 mg/kg via intravenous infusion on days -16, -3, 12, and 26; Melphalan 200 mg/m2 Ivia intravenous infusion on day -3; ASCT on day -2; ENK infusion on day 0; ALT-803 (Interleukin-15 superagonist) 10 ug/kg via subcutaneous injection on days 1, 8, 15, and 22.
  Interventions: Drug: Elotuzumab; Drug: Melphalan; Procedure: Autologous Stem Cell Transplant (ASCT); Biological: Expanded Natural Killer (ENK) Cells; Drug: ALT-803

INTERVENTIONS:
Drug: Elotuzumab — Elotuzumab 10 mg/kg via intravenous infusion on days -16, -3, 12, and 26
  Other Names: Empliciti
Drug: Melphalan — Melphalan 200 mg/m2 Ivia intravenous infusion on day -3
Procedure: Autologous Stem Cell Transplant (ASCT) — ASCT on day -2
Biological: Expanded Natural Killer (ENK) Cells — ENK cell infusion on day 0
Drug: ALT-803 — ALT-803 (Interleukin-15 superagonist) 10 ug/kg via subcutaneous injection on days 1, 8, 15, and 22
  Other Names: IL-15 superagonist

SUMMARY:
This study will evaluate the ability of Expanded Natural Killer (ENK) cells to treat multiple myeloma when administered as part of a regimen consisting of Elotuzumab and a stem cell transplant. Natural killer cells are a special type of white blood cells that are already present in the body which have the ability to kill myeloma cells. In this study, natural killer cells will be collected and then treated in a laboratory to activate and 'expand' the number of cells to increase the dose and the anti-myeloma activity of the cells before they are transfused back into the subject. Elotuzumab is a protein drug approved by the United States Food and Drug Administration (FDA) for patients with previously treated multiple myeloma and works by activating natural killer cells already present in the body and targeting a protein called SLAMF7 which is present on both natural killer cells and myeloma cells. The investigators hope that administering Elotuzumab in combination with ENK cells will enhance the anti-myeloma activity of the ENK cells.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma patients that have completed induction chemotherapy and peripheral blood stem cell collection (PBSC) in preparation for ASCT.
* Patients must have high-risk disease as defined by Gene Expression Profiling (GEP) 70 risk score of ≥ 0.66 or GEP 80 gene score of ≥ 2.48 or metaphase cytogenetic abnormalities or lactate dehydrogenase (LDH) ≥ 360 U/L (Rule out hemolysis, infection and contact PI for clarification if any doubt).
* Patients must have failed prior treatment for their multiple myeloma (MM) including a proteasome inhibitor and immunomodulatory drug (so-called 'double refractory'). Patients who have received prior salvage combination chemotherapy after failure of proteasome inhibitor and immunomodulatory drug are eligible (frank relapse at the time of enrollment is not required)
* Zubrod ≤ 2, unless solely due to symptoms of MM-related (bone) disease.
* Patients must have a platelet count of ≥ 20,000/μL within 30 days of enrollment, unless lower levels are explained by extensive bone marrow plasmacytosis or extensive prior therapy.
* Patients must be at least 18 years of age and not older than 75 years of age at the time of registration.
* must have preserved renal function as defined by a serum creatinine level of ≤ 3 mg/dL within 30 days of registration.
* Participants must have an ejection fraction by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan ≥ 40% within 90 days prior to registration.
* Patients must have adequate pulmonary function studies ≥ 50% of predicted on mechanical aspects and diffusion capacity (DLCO) ≥ 50% of predicted within 90 days prior to registration. If the patient is unable to complete pulmonary function tests due to MM-related pain or condition, exception may be granted if the principal investigator documents that the patient is a candidate for high-dose therapy.
* Patients must have at least 2x106 CD34+ cells/kg stored for transplant. In addition, there will be a 'back-up' available of 2x106 CD34+ cells/kg2x106 CD34+ cells/kg
* Patients must have signed an Institutional Review Board-approved informed consent and HIPAA authorization form.

Exclusion Criteria:

* Prior allo-transplant.
* Prior auto-transplantation is permitted provided the patient is still presently a transplant candidate and at least 2 months should have passed since last auto-transplant
* History of poorly-controlled hypertension, diabetes mellitus, or any other serious medical illness or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol or could be considered to be an exclusion criterion deemed by the PI.
* Patients must not have prior malignancy, except for adequately-treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has not received treatment for one year prior to enrollment. Other cancers will only be acceptable if the patient's life expectancy exceeds three years as determined by the PI.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy test documented within one week of registration. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* The subject may not be positive for HIV I/II or HTLV-I/II.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Multiple Myeloma Response | 98 days post-ENK infusion (100 days post-ASCT)
  Response will be measured according to International Myeloma Working Group (IMWG) Criteria

SECONDARY OUTCOMES:
Adverse Events | within 98 days post-ENK infusion (100 days post-ASCT)
  Frequency and severity of treatment-related adverse events
Persistence of ENK cells by flow cytometry and/or cytometry by time of flight (CyTOF) | within 98 days post-ENK infusion (100 days post-ASCT)

CONTACTS AND LOCATIONS:
Overall Officials: Frits van Rhee, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States